CLINICAL TRIAL: NCT01831622
Title: Influence of Stimulant Medication on Brain Processes for Decision Making in Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mats Fredriksen (Other)
Collaborators: The Research Council of Norway (Other); The Hospital of Vestfold (Other); Norwegian Institute of Public Health (Other Government)
Responsible Party: Sponsor-Investigator, Mats Fredriksen, Researcher MD, PhD, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012-005246-38; 2012-005246-38 (EudraCT Number); 2012/1105-8 (Other: Regional Ethics Commitees); 2011/1585-10 (Other: Regional Ethics Commitees)
Record Dates: First submitted 2013-04-09; First posted 2013-04-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Attention Deficit-Hyperactivity Disorder
Keywords: Decision-Making; functional MRI; pharmacological MRI; Reinforcement Learning; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; 5,10-dihydro-5-methylphenazine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral (Experimental): Cognitive testing of participants. Asterisk applies for patient group.
  Day 1:
  * Patient arrives having abstained medication for minimum 20 hours.*
  * Administer either Ritalin or placebo intervention, and wait 60 minutes before computer-testing.*
  * Case Report Form (CRF), ASRS and Wechsler Adult Intelligence Scale (WAIS) subtests.
  * Blood sample, if consented.*
  * Computerized testing.
  * Administer opposite treatment.*
  Day 2:
  * Patient arrives having abstained medication for a minimum of 20 hours.*
  * Administer either Ritalin or placebo intervention (opposite of Day 1), and wait 60 minutes before computer-testing.*
  * CRF 3, ASRS and Edinburgh Handedness Inventory (EHI).
  * Blood sample, if consented.*
  * Computerized testing.
  * Administer opposite treatment.*
  Interventions: Drug: Ritalin; Drug: Placebo
- fMRI-arm (Experimental): Asterisk applies only for patient group.
  Day 1:
  * Patient arrives having abstained medication for minimum 20 hours.*
  * Administer either Ritalin or placebo intervention, and wait 60 minutes before MRI testing.*
  * CRF 2, Adult ASRS and WAIS subtests.
  * Blood sample, if consented.*
  * Computerized testing.
  * Administer opposite treatment to ensure the patients have not been withheld from medication for too long while keeping blind.*
  Day 2 (after 14 - 40 days):
  * Patient arrives having abstained medication for a minimum of 20 hours.*
  * Administer either Ritalin or placebo intervention, and wait 60 minutes before testing (opposite of Day 1).*
  * CRF 3, ASRS and EHI.
  * Blood sample, if consented.*
  * Computerized testing.
  * Administer opposite treatment.*
  Interventions: Drug: Ritalin; Drug: Placebo

INTERVENTIONS:
Drug: Ritalin — On one of the two test-dates the patient participant is administered methylphenidate, in the dose prescribed by the patients doctor.
  Other Names: Methylphenidate; MPH
Drug: Placebo — On one of the test-dates the patient participants are administered a sugar pill, matching their prescribes medical dose.
  Other Names: Sugar pill

SUMMARY:
The goal of this trial is to investigate the cognitive- and brain-mechanisms underlying decision making (DM) and learning in young adults with Attention-Deficit/Hyperactivity Disorder (ADHD) as well as the modulation of task-related and task-independent brain activation by methylphenidate. The study aims at using a double-blinded, placebo controlled, cross-over, withdrawal design to study the effects of ADHD and methylphenidate in both a behavioural study investigating cognitive effects on decision making and instrumental learning, and a functional MRI (fMRI) study investigating the effects on brain mechanisms during decision making alone. A secondary objective of the trial is to measure the effect of adult ADHD and methylphenidate on cerebral perfusion. This will be done through applying a novel arterial spin labelling MRI-technique on the participants in the fMRI arm of the study.

DETAILED DESCRIPTION:
The immediate scientific goal of this trial is to investigate the cognitive- and brain-mechanisms underlying Decision Making (DM) and instrumental learning in young adults with ADHD as well as the modulation of task-related and task-independent brain activation by MPH. In a more applied perspective, the investigators hope this trial will contribute to the development of tools for improved diagnosis and treatment monitoring of ADHD. Diagnostic tools should be based on the understanding of cognitive and brain mechanisms contributing to the symptom manifestation of ADHD. The study aims at using a double-blinded, placebo controlled cross-over withdrawal design to study the effects of ADHD and MPH in both a behavioural study investigating cognitive effects on DM and instrumental learning, and an fMRI study investigating the effects on brain mechanisms during DM alone. The results of the behavioural DM task from the fMRI experiment will be pooled with the data from the behavioural study to achieve higher statistical power in the analysis of the behavioural data.

A distinctive characteristic of this proposal is to gain insight into differences between ADHD-patients and healthy controls and the effects of methylphenidate (MPH) medication with an approach termed "computational psychiatry" (Maia and Frank, 2011). In this approach, the investigators apply mathematical models of cognition to observed behaviour in order to derive latent decision variables characterizing the DM- and instrumental learning processes. When combined with neuroimaging methods, computational models allow identification of differences in affective and cognitive processes together with the neurobiological processes that underlie these differences (Frank et al., 2004). Such insights should be the foundation of new tools for diagnosis and therapeutic treatment of ADHD.

ELIGIBILITY:
Inclusion Criteria:

Drug-Naïve Group

* Comply with Diagnostic and Statistical Manual (DSM) -IV criteria for ADHD.
* No history of medication with Methylphenidate.
* Must be between the age of 18 and 40.
* Signed informed consent and expected cooperation of the patients for the intervention and the test dates must be obtained and documented according to International Conference on Harmonisation (ICH) Good Clinical Practice (GCP), and national/local regulations.
* After stable medication is established, these will be incorporated into the study following the procedures of the "drug group".

Drug group

* Comply with DSM-IV criteria for ADHD.
* On stable treatment with MPH.
* Must be between the age of 18 and 40.
* Signed informed consent and expected cooperation of the patients for the intervention and the test dates must be obtained and documented according to ICH GCP, and national/local regulations.

Healthy Control Group

* Must be between the age of 18 and 40.
* No current psychiatric diagnosis.
* Signed informed consent and expected cooperation of the patients for the intervention and the test dates must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

* Treatment with the following groups of pharmacological agents will be considered as exclusion criteria for participation:
* Antidepressants (MOA-inhibitors, Tricyclic antidepressants, Selective Serotonin Re-uptake Inhibitors)
* Antipsychotics (both first and second generation)
* Anxiolytics/hypnotics (benzodiazepines, barbiturates)
* Opiates
* History of alcohol or drug abuse.
* History of moderate to severe head injury.
* Major psychiatric comorbidity (i.e. psychosis, active suicidal ideation or acute exacerbation of other psychiatric condition in need of immediate treatment).
* Epilepsy
* History of severe memory loss
* Under treatment for metabolic disorders
* Severe primary sensory loss
* Any condition contraindicating treatment with methylphenidate will automatically lead to exclusion, since these patients will not receive methylphenidate from clinician and thus will not meet inclusion criteria (including pregnancy, methylphenidate allergies, incompatible concomitant medication etc.).
* MRI specific criteria: contraindications for MRI (i.e. metallic or circuit-containing implants, severe claustrophobia)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Effect of ADHD medication on decision making | by may 2015 (up to 3 years)
  The study will both use standard statistical models on reaction time and accuracy data, but also use Bayesian Statistics and mathematical modelling.
  The investigators expect higher Drift Diffusion Model drift rate in the controls and patients on medication, and slower drift rate for participants off medication.

CONTACTS AND LOCATIONS:
Overall Officials: Mats Fredriksen, MD, Principal Investigator — Vestre Viken Hospital Trust and the University of Oslo; Guido P Biele, PhD, Study Director — University of Oslo; Tor Endestad, PhD, Study Chair — University of Oslo
Locations (2):
- Norway (2):
  - Department of Psychology, University of Oslo, Oslo, Oslo County
  - Adult ADHD diagnostic clinic, Vestre Viken Hospital Trust, Tønsberg, Tønsberg

REFERENCES:
- [Derived] Mowinckel AM, Alnaes D, Pedersen ML, Ziegler S, Fredriksen M, Kaufmann T, Sonuga-Barke E, Endestad T, Westlye LT, Biele G. Increased default-mode variability is related to reduced task-performance and is evident in adults with ADHD. Neuroimage Clin. 2017 Mar 30;16:369-382. doi: 10.1016/j.nicl.2017.03.008. eCollection 2017. PMID 28861338